CLINICAL TRIAL: NCT02097745
Title: An Open Label Study of the Efficacy and Safety of Re-treatments With Rituximab (MabThera/Rituxan) in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Anti-TNFa Therapies
Brief Title: A Study of the Efficacy and Safety of Re-treatments With Rituximab in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Anti-tnfa Therapies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WA17531; NCT00468377 (obsolete NCT alias)
Record Dates: First submitted 2014-03-20; First posted 2014-03-27 (Estimated); Results first posted 2014-11-07 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Rituximab

ARMS (1):
- MabThera/Rituxan (Experimental)
  Interventions: Drug: methotrexate; Drug: rituximab [MabThera/Rituxan]

INTERVENTIONS:
Drug: methotrexate — a 10-25 mg stable dose given orally or parenterally throughout study
Drug: rituximab [MabThera/Rituxan] — 1 g given by intravenous infusion on Days 1 and 15 of each treatment course
  Other Names: MabThera/Rituxan

SUMMARY:
This study will assess the long-term safety and efficacy of repeating treatment with MabThera, in combination with methotrexate and steroids, in patients who were previously randomized into MabThera study WA17042. The anticipated time on study treatment is until Mabthera is available on the local market and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 18-80 years of age with active RA;
* patients who participated in MabThera study WA17042, and completed to at least the Week 24 visit;
* eligible for re-treatment, based on clinical symptoms;
* patients of reproductive potential must be using reliable contraceptive methods.

Exclusion Criteria:

* patients who participated in MabThera study WA17042 but withdrew into the safety follow-up;
* current treatment with any other disease-modifying antirheumatic drug (apart from methotrexate), or any anti-TNFalfa, anti-IL1, or other biologic therapies;
* development of any new contraindications to receiving MabThera;
* women who are pregnant or breast-feeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2004-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (86):
- United States (50):
  - Mesa, Arizona
  - Paradise Valley, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Fullerton, California
  - Los Angeles, California
  - Pasadena, California
  - Rancho Mirage, California
  - Santa Maria, California
  - Danbury, Connecticut
  - Boca Raton, Florida
  - Delray Beach, Florida
  - Fort Lauderdale, Florida
  - Jupiter, Florida
  - Orlando, Florida
  - Boise, Idaho
  - Coeur d'Alene, Idaho
  - Meridian, Idaho
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Shreverport, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Albany, New York
  - Manhasset, New York
  - New York, New York
  - Rochester, New York
  - Smithtown, New York
  - Chapel Hill, North Carolina
  - Greenville, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Mayfield, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Amarillo, Texas
  - Dallas, Texas
  - Houston, Texas
  - Waco, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Seattle, Washington
  - Spokane, Washington
  - Madison, Wisconsin
- Belgium (2):
  - Brussels
  - Ghent
- Canada (5):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
- France (5):
  - Bois-Guillaume
  - Le Kremlin-Bicêtre
  - Montpellier
  - Paris
  - Toulouse
- Germany (5):
  - Berlin
  - Dresden
  - Leipzig
  - Ratingen
  - Würzburg
- Ireland (2):
  - Cork
  - Dublin
- Israel (5):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Italy (3):
  - Udine, Friuli Venezia Giulia
  - Brescia, Lombardy
  - Pisa, Tuscany
- Amsterdam, Netherlands
- Norway (3):
  - Drammen
  - Oslo
  - Tromsø
- United Kingdom (5):
  - Cannock
  - Leeds
  - London
  - Manchester
  - Newcastle upon Tyne

REFERENCES:
- [Derived] Keystone E, Fleischmann R, Emery P, Furst DE, van Vollenhoven R, Bathon J, Dougados M, Baldassare A, Ferraccioli G, Chubick A, Udell J, Cravets MW, Agarwal S, Cooper S, Magrini F. Safety and efficacy of additional courses of rituximab in patients with active rheumatoid arthritis: an open-label extension analysis. Arthritis Rheum. 2007 Dec;56(12):3896-908. doi: 10.1002/art.23059. PMID 18050221

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab: Participants received rituximab 1 g intravenously (IV) on Days 1 and 15 of each course of retreatment. In addition, participants received methotrexate 10-25 mg/week orally or parenterally, methylprednisolone 100 mg IV 30 minutes prior to both rituximab infusions, and a stable dose of folic acid ≥ 5 mg/week or equivalent, given as either a single dose or as divided daily doses.
Period: Overall Study
Arm/Group | Rituximab
Started | 335 (Six participants did not receive any treatment and were not included in any analyses.)
Completed | 157
Not Completed | 178
Not completed — Adverse Event | 25
Not completed — Death | 16
Not completed — Failure to Return | 14
Not completed — Administrative/Other | 27
Not completed — Reason Not Specified | 96

BASELINE CHARACTERISTICS:
Population: Safety population: All participants who received any part of an infusion of study medication.
Arm/Group | Rituximab
Number analyzed (Participants) | 335
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 273
  Male | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20 (ACR20) Response
Description: A patient had an ACR20 response if there was at least a 20% improvement, ie, reduction from Baseline, in tender and swollen joint counts (28 assessed joints) and in at least 3 of the following 5 parameters: Separate patient and physician assessments of patient disease activity in the previous 24 hours on a visual analog scale (VAS, left end=no disease activity [symptom-free and no arthritis symptoms], right end=maximum disease activity; patient assessment of pain in previous 24 hours on a VAS (left end=no pain and right end=unbearable pain); Health Assessment Questionnaire-Disability Index (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do); and acute-phase reactant (either C-reactive protein or erythrocyte sedimentation rate). The ACR20 response was compared to Baseline in the precursor study WA17042. The first retreatment may have occurred in the precursor study WA17042.
Time Frame: Baseline to the end of the retreatment period (up to 7 years, 6 months)
Population: Intent-to-treat population: All participants who received any part of an infusion of study medication in study WA17531.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 335
Percentage of participants
  Retreatment 1 (n = 320) | 67.5
  Retreatment 2 (n = 267) | 74.9
  Retreatment 3 (n = 234) | 73.9
  Retreatment 4 (n = 175) | 67.4
  Retreatment 5 (n = 136) | 69.9
  Retreatment 6 (n = 92) | 72.8

2. Secondary Outcome: Change From Baseline in the Disease Activity Score 28 (DAS28)
Description: The DAS28 is an index for measuring disease activity in rheumatic arthritis and includes swollen and tender joint counts, erythrocyte sedimentation rate (ESR), and general health (GH) status. The index is calculated with the following formula: DAS28 = (0.56 × √(TJC28)) + (0.28 × √(SJC28)) + (0.7 × log(ESR)) + (0.014 × GH), where TJC28 = tender joint count and SJC28 = swollen joint count, each on 28 joints. GH = a patient's global assessment of disease activity in the previous 24 hours on a 100 mm visual analog scale (left end = no disease activity [symptom-free and no arthritis symptoms], right end = maximum disease activity [maximum arthritis disease activity]). When ESR equaled 0 mm/hr, it was set to 1 mm/hr. The DAS28 scale ranges from 0 to 10, where a higher score represents higher disease activity. A negative change score indicates improvement. The first retreatment may have occurred in the precursor study WA17042.
Time Frame: Baseline to the end of the retreatment period (up to 7 years, 6 months)
Population: Intent-to-treat population: All participants who received any part of an infusion of study medication in study WA17531.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 335
Units on a scale
  Retreatment 1 (n = 304) | -2.32 (1.336)
  Retreatment 2 (n = 258) | -2.77 (1.302)
  Retreatment 3 (n = 227) | -3.01 (1.388)
  Retreatment 4 (n = 168) | -3.05 (1.537)
  Retreatment 5 (n = 132) | -3.15 (1.536)
  Retreatment 6 (n = 87) | -2.96 (1.540)

3. Secondary Outcome: Percentage of Participants With DAS28 Low Disease Activity and DAS28 Remission
Description: The DAS28 is an index for measuring disease activity in rheumatic arthritis and includes swollen and tender joint counts, erythrocyte sedimentation rate (ESR), and general health (GH) status. The index is calculated with the following formula: DAS28 = (0.56 × √(TJC28)) + (0.28 × √(SJC28)) + (0.7 × log(ESR)) + (0.014 × GH), where TJC28 = tender joint count and SJC28 = swollen joint count, each on 28 joints. GH = a patient's global assessment of disease activity in the previous 24 hours on a 100 mm visual analog scale (left end = no disease activity [symptom-free and no arthritis symptoms], right end = maximum disease activity [maximum arthritis disease activity]). When ESR equaled 0 mm/hr, it was set to 1 mm/hr. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. Low disease activity was defined as a DAS28 score ≤ 3.2. DAS28 remission was defined as a DAS28 score < 2.6. The first retreatment may have occurred in the precursor study WA17042.
Time Frame: Baseline to the end of the retreatment period (up to 7 years, 6 months)
Population: Intent-to-treat population: All participants who received any part of an infusion of study medication in study WA17531.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 335
Percentage of participants
  Retreatment 1: Low Disease Activity (n=314) | 17.2
  Retreatment 1: Remission | 8.9
  Retreatment 2: Low Disease Activity (n=265) | 27.9
  Retreatment 2: Remission | 15.1
  Retreatment 3: Low Disease Activity (n=234) | 36.8
  Retreatment 3: Remission | 18.8
  Retreatment 4: Low Disease Activity (n=172) | 33.7
  Retreatment 4: Remission | 20.9
  Retreatment 5: Low Disease Activity (n=135) | 36.3
  Retreatment 5: Remission | 20.0
  Retreatment 6: Low Disease Activity (n=90) | 33.3
  Retreatment 6: Remission | 15.6

4. Secondary Outcome: Percentage of Participants With Good, Moderate, or no European League Against Rheumatism (EULAR) Responses
Description: Change of the Disease Activity Score 28 score from baseline was used to determine EULAR responses of good, moderate, or no response. For a post-baseline score ≤ 3.2, a change from baseline of < -1.2 was a good response, < -0.6 to ≥ -1.2 was a moderate response, and ≥ -0.6 was no response. For a post-baseline score > 3.2 to ≤ 5.1, a change from baseline of < -0.6 was a moderate response and ≥ -0.6 was no response. For a post-baseline score > 5.1, a change from baseline < -1.2 was a moderate response and ≥ -1.2 was no response. A good response could not be achieved for post-baseline scores > 3.2. The first retreatment may have occurred in the precursor study WA17042.
Time Frame: Baseline to the end of the retreatment period (up to 7 years, 6 months)
Population: Intent-to-treat population: All participants who received any part of an infusion of study medication in study WA17531.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 335
Percentage of participants
  Retreatment 1: Good Response (n = 304) | 17.1
  Retreatment 1: Moderate Response | 64.8
  Retreatment 1: No Response | 18.1
  Retreatment 2: Good Response (n = 258) | 27.5
  Retreatment 2: Moderate Response | 64.3
  Retreatment 2: No Response | 8.1
  Retreatment 3: Good Response (n = 227) | 36.6
  Retreatment 3: Moderate Response | 53.3
  Retreatment 3: No Response | 10.1
  Retreatment 4: Good Response (n = 168) | 33.9
  Retreatment 4: Moderate Response | 58.9
  Retreatment 4: No Response | 7.1
  Retreatment 5: Good Response (n = 132) | 36.4
  Retreatment 5: Moderate Response | 54.5
  Retreatment 5: No Response | 9.1
  Retreatment 6: Good Response (n = 87) | 33.3
  Retreatment 6: Moderate Response | 59.8
  Retreatment 6: No Response | 6.9

5. Secondary Outcome: Change From Baseline in the American College of Rheumatology n (ACRn) Response
Description: The ACRn response was defined as each participant's least favorable percentage change from Baseline in 3 measures, tender joint count, swollen joint count (28 assessed joints), and improvement score achieved in at least 3 of the 5 remaining ACR parameters: Separate patient and physician assessments of patient disease activity in the previous 24 hours on a visual analog scale (VAS, left end=no disease activity, right end=maximum disease activity; patient assessment of pain in previous 24 hours on a VAS (left end=no pain, right end=unbearable pain); Health Assessment Questionnaire-Disability Index (20 questions, 8 components, 0=without difficulty to 3=unable to do); and acute-phase reactant (either C-reactive protein or erythrocyte sedimentation rate). A higher change percentage indicates greater improvement from Baseline. The ACRn response was compared to Baseline in the precursor study WA17042. The first retreatment may have occurred in the precursor study WA17042.
Time Frame: Baseline to the end of the retreatment period (up to 7 years, 6 months)
Population: Intent-to-treat population: All participants who received any part of an infusion of study medication in study WA17531.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Rituximab
Number analyzed (Participants) | 335
Percentage change
  Retreatment 1 (n = 320) | 32.04 (37.709)
  Retreatment 2 (n = 267) | 39.25 (35.494)
  Retreatment 3 (n = 234) | 39.89 (41.166)
  Retreatment 4 (n = 175) | 37.71 (43.201)
  Retreatment 5 (n = 136) | 37.59 (41.109)
  Retreatment 6 (n = 92) | 35.53 (38.650)

6. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: The HAQ-DI is a questionnaire specific for rheumatoid arthritis and consists of 20 questions referring to 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Participants completed the questionnaire by answering the 20 questions on a scale of 0 (without difficulty) to 3 (unable to do). The total score ranges from 0 (no disability) to 3 (completely disabled). A negative change score indicates improvement.
Time Frame: Baseline to the end of the retreatment period (up to 7 years, 6 months)
Population: Intent-to-treat population: All participants who received any part of an infusion of study medication in study WA17531.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 335
Units on a scale
  Retreatment 1 (n = 320) | -0.51 (0.569)
  Retreatment 2 (n = 267) | -0.54 (0.569)
  Retreatment 3 (n = 234) | -0.56 (0.601)
  Retreatment 4 (n = 175) | -0.55 (0.603)
  Retreatment 5 (n = 136) | -0.60 (0.647)
  Retreatment 6 (n = 92) | -0.55 (0.653)

7. Secondary Outcome: Change From Baseline in the Physical and Mental Component Scores of the Short Form 36 (SF-36) Health Survey
Description: The SF-36 Health Survey uses patient-reported symptoms on 8 subscales to assess health-related quality of life (HRQoL). The Physical Component Summary (PCS) score summarizes the subscales Physical Functioning, Role-Physical, Bodily Pain, and General Health. The Mental Component Summary (MCS) score summarizes the subscales Vitality, Social Functioning, Role-Emotional, and Mental Health. Each score was scaled from 0 to 100 with a higher score indicating better HRQoL. A positive change score indicates an improvement in HRQoL.
Time Frame: Baseline to the end of the retreatment period (up to 7 years, 6 months)
Population: Intent-to-treat population: All participants who received any part of an infusion of study medication in study WA17531.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 335
Units on a scale
  Retreatment 1: Physical Health (n = 249) | 7.383 (8.4618)
  Retreatment 1: Mental Health | 5.550 (12.0705)
  Retreatment 2: Physical Health (n = 255) | 6.018 (7.9757)
  Retreatment 2: Mental Health | 5.746 (10.7778)
  Retreatment 3: Physical Health (n = 220) | 6.206 (8.2326)
  Retreatment 3: Mental Health | 4.777 (10.1916)
  Retreatment 4: Physical Health (n = 167) | 5.660 (7.9137)
  Retreatment 4: Mental Health | 4.864 (10.2215)
  Retreatment 5: Physical Health (n = 124) | 5.038 (8.2643)
  Retreatment 5: Mental Health | 5.141 (11.8848)
  Retreatment 6: Physical Health (n = 88) | 5.214 (7.5370)
  Retreatment 6: Mental Health | 2.658 (9.8556)

8. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Score
Description: The FACIT-F is a 13-item participant self-reporting questionnaire that assesses fatigue over the previous 7 days by scoring each item on a 5-point scale (0=Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit, 4=Very much). An overall FACIT-F score was obtained by summing the scores of all 13 items. The overall score ranged from 0 to 52. A lower score indicates less fatigue. A negative change score indicates improvement.
Time Frame: Baseline to the end of the retreatment period (up to 7 years, 6 months)
Population: Intent-to-treat population: All participants who received any part of an infusion of study medication in study WA17531.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 335
Units on a scale
  Retreatment 1 (n = 321) | 10.790 (10.7934)
  Retreatment 2 (n = 272) | 6.390 (9.1312)
  Retreatment 3 (n = 232) | 7.075 (9.8208)
  Retreatment 4 (n = 176) | 6.770 (10.4043)
  Retreatment 5 (n = 131) | 8.030 (10.4571)
  Retreatment 6 (n = 89) | 5.429 (9.4251)

9. Secondary Outcome: Percentage of Participants With no Radiographic Progression From Baseline to Year 5
Description: Radiographic progression was defined as a change of ≤ 0 in the total Genant-modified Sharp score. The Genant-modified Sharp scoring system assesses structural damage due to rheumatoid arthritis in radiographs. A score for erosions of 0-3.5 (8 gradations) is assigned for 14 joints in each hand and wrist, and 6 joints in each foot. Joint space narrowing scores of 0-4 (9 gradations) are assigned to 13 joints in each hand and 6 joints in each foot. The maximum erosion score is 40 x 3.5 = 140. The maximum joint space narrowing score is 38 x 4.0 = 152. Both the erosion and joint space narrowing scores are normalized to 145 and are added together for a maximum total Genant-modified Sharp score of 290; the minimum score is 0. A higher score indicates more damage. Data is reported for 2 groups.
Time Frame: Baseline to Year 5
Population: Intent-to-treat population: All participants who received any part of an infusion of study medication in study WA17531. Only participants who had radiographs available at Baseline and Year 5 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Placebo: Data for participants who received placebo in study WA17042 are included in this reporting group for data collected up until they received their first dose of rituximab in this study (study WA17531). Data from these participants collected after the first dose of rituximab are included in the rituximab reporting group.
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 79 | 105
Percentage of participants | 21.5 [12.0 to 31.0] | 32.4 [23.0 to 41.0]

10. Secondary Outcome: Change From Baseline in the Total Genant-modified Sharp Score at Year 5
Description: The Genant-modified Sharp scoring system assesses structural damage due to rheumatoid arthritis in radiographs. A score for erosions of 0-3.5 (8 gradations) is assigned for 14 joints in each hand and wrist, and 6 joints in each foot. Joint space narrowing scores of 0-4 (9 gradations) are assigned to 13 joints in each hand and 6 joints in each foot. The maximum erosion score is 40 x 3.5 = 140. The maximum joint space narrowing score is 38 x 4.0 = 152. Both the erosion and joint space narrowing scores are normalized to 145 and are added together for a maximum total Genant-modified Sharp score of 290; the minimum score is 0. A higher score indicates more damage. A negative change score indicates improvement. Data is reported for 2 groups.
Time Frame: Baseline to Year 5
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 79 | 105
Units on a scale | 5.446 (8.4701) | 3.202 (6.5538)

11. Secondary Outcome: Change From Baseline in the Genant-modified Sharp Erosion Score at Year 5
Description: The Genant-modified Sharp scoring system assesses structural damage due to rheumatoid arthritis in radiographs. A score for erosions of 0-3.5 (8 gradations) is assigned for 14 joints in each hand and wrist, and 6 joints in each foot. The maximum erosion score is 40 x 3.5 = 140 which is normalized to 145. The minimum score is 0 and the maximum score is 145. A higher score indicates more damage. A negative change score indicates improvement. Data is reported for 2 groups.
Time Frame: Baseline to Year 5
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 79 | 105
Units on a scale | 3.101 (4.8980) | 1.880 (4.4491)

12. Secondary Outcome: Change From Baseline in the Genant-modified Sharp Joint Space Narrowing Score at Year 5
Description: The Genant-modified Sharp scoring system assesses structural damage due to rheumatoid arthritis in radiographs. A score joint space narrowing of 0-4 (9 gradations) is assigned to 13 joints in each hand and 6 joints in each foot. The maximum joint space narrowing score is 38 x 4.0 = 152 which is normalized to a score of 145. The minimum score is 0 and the maximum score is 145. A higher score indicates more damage. A negative change score indicates improvement. Data is reported for 2 groups.
Time Frame: Baseline to Year 5
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 79 | 105
Units on a scale | 2.344 (4.3263) | 1.322 (2.7831)

13. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Year 5
Description: The HAQ-DI is a questionnaire specific for rheumatoid arthritis and consists of 20 questions referring to 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Participants completed the questionnaire by answering the 20 questions on a scale of 0 (without difficulty) to 3 (unable to do). The total score ranges from 0 (no disability) to 3 (completely disabled). A negative change score indicates improvement. Data is reported for 2 groups.
Time Frame: Baseline to Year 5
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 75 | 100
Units on a scale | -0.408 (0.5348) | -0.540 (0.6521)

ADVERSE EVENTS:
Description: Safety population: All participants who received any part of an infusion of study medication in this study.
Arm/Group | Placebo | Rituximab
Serious Adverse Events (participants affected / at risk) | 14/140 | 197/335
Other Adverse Events (participants affected / at risk) | 112/140 | 327/335
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=140) | Rituximab (N=335)
Pneumonia (Infections and infestations) | 0 | 10
Cellulitis (Infections and infestations) | 0 | 6
Gastroenteritis (Infections and infestations) | 0 | 4
Pyelonephritis (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 0 | 4
Bronchitis (Infections and infestations) | 0 | 3
Bronchopneumonia (Infections and infestations) | 0 | 3
Escherichia urinary tract infection (Infections and infestations) | 0 | 3
Appendicitis (Infections and infestations) | 0 | 2
Arthritis infective (Infections and infestations) | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 2
Pneumonia streptococcal (Infections and infestations) | 0 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 2
Abdominal wall abscess (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess intestinal (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cytomegalovirus duodenitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Muscle abscess (Infections and infestations) | 0 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Post procedural cellulitis (Infections and infestations) | 0 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Salmonella sepsis (Infections and infestations) | 0 | 1
Scedosporium infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Shigella infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal abscess (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Zoonosis (Infections and infestations) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 23
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 10
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Hand deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint instability (Metabolism and nutrition disorders) | 0 | 1
Ligament calcification (Musculoskeletal and connective tissue disorders) | 0 | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 5
Myocardial infarction (Cardiac disorders) | 1 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 4
Angina pectoris (Cardiac disorders) | 0 | 3
Pericarditis (Cardiac disorders) | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 2
Sick sinus syndrome (Cardiac disorders) | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 13
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 4
Accident (Injury, poisoning and procedural complications) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Large intestine perforation (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Diverticular perforation (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2
Umbilical hernia (Gastrointestinal disorders) | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Protein-losing gastroenteropathy (Gastrointestinal disorders) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Infusion related reaction (General disorders) | 0 | 5
Pyrexia (General disorders) | 0 | 4
Surgical failure (General disorders) | 0 | 3
Chest pain (General disorders) | 0 | 2
Device failure (General disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Device breakage (General disorders) | 0 | 1
Device dislocation (General disorders) | 0 | 1
Device occlusion (General disorders) | 0 | 1
Inflammation (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 4
Transient ischaemic attack (Nervous system disorders) | 0 | 3
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cluster headache (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 2
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Aortic occlusion (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Arterial haemorrhage (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Poor peripheral circulation (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Diabetic complication (Metabolism and nutrition disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 1
Urogenital prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 4
Major depression (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Eosinophilic cystitis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Respiratory rate decreased (Investigations) | 0 | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Physical assault (Social circumstances) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=140) | Rituximab (N=335)
Upper respiratory tract infection (Infections and infestations) | 14 | 132
Nasopharyngitis (Infections and infestations) | 12 | 101
Urinary tract infection (Infections and infestations) | 11 | 86
Bronchitis (Infections and infestations) | 9 | 81
Sinusitis (Infections and infestations) | 13 | 68
Gastroenteritis (Infections and infestations) | 2 | 48
Gastroenteritis viral (Infections and infestations) | 2 | 45
Influenza (Infections and infestations) | 2 | 42
Cellulitis (Infections and infestations) | 1 | 25
Rhinitis (Infections and infestations) | 3 | 22
Tooth abscess (Infections and infestations) | 1 | 23
Oral herpes (Infections and infestations) | 4 | 19
Pneumonia (Infections and infestations) | 2 | 21
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 22
Ear infection (Infections and infestations) | 1 | 19
Herpes zoster (Infections and infestations) | 3 | 17
Pharyngitis (Infections and infestations) | 0 | 20
Oral candidiasis (Infections and infestations) | 0 | 17
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 57 | 217
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 68
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 47
Bursitis (Musculoskeletal and connective tissue disorders) | 3 | 38
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 30
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 31
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 21
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 22
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 22
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 19
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 18
Infusion related reaction (General disorders) | 26 | 155
Fatigue (General disorders) | 4 | 40
Oedema peripheral (General disorders) | 1 | 43
Pyrexia (General disorders) | 3 | 20
Influenza like illness (General disorders) | 1 | 17
Nausea (Gastrointestinal disorders) | 8 | 55
Diarrhoea (Gastrointestinal disorders) | 12 | 45
Vomiting (Gastrointestinal disorders) | 3 | 31
Abdominal pain (Gastrointestinal disorders) | 6 | 24
Constipation (Gastrointestinal disorders) | 3 | 25
Dyspepsia (Gastrointestinal disorders) | 0 | 26
Abdominal pain upper (Gastrointestinal disorders) | 2 | 19
Dental caries (Gastrointestinal disorders) | 1 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 50
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 22
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 23
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 19
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 19
Depression (Psychiatric disorders) | 5 | 52
Insomnia (Psychiatric disorders) | 5 | 40
Anxiety (Psychiatric disorders) | 1 | 18
Headache (Nervous system disorders) | 7 | 61
Dizziness (Nervous system disorders) | 2 | 25
Paraesthesia (Nervous system disorders) | 0 | 18
Rash (Skin and subcutaneous tissue disorders) | 8 | 49
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 18
Fall (Injury, poisoning and procedural complications) | 4 | 71
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 35
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 25
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 18
Hypertension (Vascular disorders) | 4 | 58
Cataract (Eye disorders) | 1 | 22
Conjunctivitis (Eye disorders) | 0 | 19
Anaemia (Blood and lymphatic system disorders) | 3 | 25
Seasonal allergy (Immune system disorders) | 2 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.